CLINICAL TRIAL: NCT01864148
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Dose-Ranging Study to Assess the Efficacy, Safety, Tolerability, and Pharmacokinetics of BIIB033 in Subjects With Relapsing Forms of Multiple Sclerosis When Used Concurrently With Avonex
Brief Title: Study to Assess the Efficacy, Safety, Tolerability, and Pharmacokinetics of BIIB033 in Participants With Relapsing Forms of Multiple Sclerosis When Used Concurrently With Avonex
Acronym: SYNERGY
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 215MS201; 2011-006262-40 (EudraCT Number)
Record Dates: First submitted 2013-05-24; First posted 2013-05-29 (Estimated); Results first posted 2017-05-03 (Actual); Last update posted 2017-05-03 (Actual); Status verified 2017-03

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — opicinumab; Interferon beta-1a

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- BIIB033, 3 mg/kg (Experimental): BIIB033 3 mg/kg once every 4 weeks intravenous (IV) infusion up to Week 72.
  Avonex once-weekly intramuscular (IM) injection up to Week 84.
  Interventions: Drug: BIIB033; Drug: Avonex
- BIIB033, 10 mg/kg (Experimental): BIIB033 10 mg/kg once every 4 weeks IV infusion up to Week 72.
  Avonex once-weekly IM injection up to Week 84.
  Interventions: Drug: BIIB033; Drug: Avonex
- BIIB033, 30 mg/kg (Experimental): BIIB033 30 mg/kg once every 4 weeks IV infusion up to Week 72.
  Avonex once-weekly IM injection up to Week 84.
  Interventions: Drug: BIIB033; Drug: Avonex
- BIIB033, 100 mg/kg (Experimental): BIIB033 100 mg/kg once every 4 weeks IV infusion up to Week 72.
  Avonex once-weekly IM injection up to Week 84.
  Interventions: Drug: BIIB033; Drug: Avonex
- Placebo (Placebo Comparator): Placebo once every 4 weeks IV infusion up to Week 72.
  Avonex once-weekly IM injection up to Week 84.
  Interventions: Other: Placebo; Drug: Avonex

INTERVENTIONS:
Drug: BIIB033
  Other Names: anti-LINGO-1 mAb
  Arms: BIIB033, 10 mg/kg; BIIB033, 100 mg/kg; BIIB033, 3 mg/kg; BIIB033, 30 mg/kg
Other: Placebo
  Arms: Placebo
Drug: Avonex
  Other Names: interferon beta-1a

SUMMARY:
The primary objective of the study is to evaluate the efficacy of BIIB033 in participants with active relapsing multiple sclerosis (MS) when used concurrently with Avonex.

Secondary objectives of this study in this study population are to assess the safety, tolerability, and population pharmacokinetics of BIIB033 when used concurrently with Avonex.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of relapsing remitting MS (RRMS) or onset of secondary progressive MS (SPMS)
* RRMS and SPMS subjects must have evidence of ongoing disease activity within 12 months of enrollment.
* All male and female subjects of childbearing potential must practice effective contraception during the study and be willing and able to continue contraception for at least 6 months after their last dose of study treatment

Key Exclusion Criteria:

* A MS relapse that has occurred within the 90 days prior to Day 1/Baseline and/or the subject has not stabilized from a previous relapse prior to Screening
* Previous history of clinically significant disease.
* Plans to undergo elective major procedures/surgeries at any time during the study.
* Treatment with any investigational MS drugs within 3 weeks or 5 times the half life (whichever is longer) prior to Day 1/Baseline
* RRMS subjects with any history of inadequate response to any approved interferon β preparation
* History of human immunodeficiency virus (HIV), hepatitis C virus antibody, or hepatitis B virus
* History or evidence of drug or alcohol abuse within 2 years prior to randomization

Note: Other protocol defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 58 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 419 (Actual)
Dates: Start 2013-08; Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (72):
- United States (11):
  - North Central Neurology Assoc PC, Cullman, Alabama
  - Phoenix Neurological Associates, Phoenix, Arizona
  - Raleigh Neurology Associates PA, Raleigh, California
  - Stanford University Medical Center, Stanford, California
  - Immunoe International Research Center, Centennial, Colorado
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Michigan Institute For Neurological Disorders, Farmington Hills, Michigan
  - Washington University, St Louis, Missouri
  - Multiple Sclerosis Center of North Eastern New York, Latham, New York
  - OMRF Multiple Sclerosis Center of Excellence, Oklahoma City, Oklahoma
  - Swedish Medical Center, Seattle, Washington
- Canada (6):
  - Research Site, Ottowa, Ontario
  - Research Site, Gatinueau, Quebec
  - Research Site, Greenfield Park, Quebec
  - Research Site, Lévis, Quebec
  - Research Site, Montreal, Quebec
  - London Health Sciences Centre, London
- Czechia (6):
  - Vseobecna Fakultni Nemocnice V Praze, Prague, Hlavní Mesto
  - Nemocnice Jihlava Prispevkova Organizace, Jihlava, Kraj Vysočina
  - Fakultni Nemocnice Hradec Kralove, Hradec Králové, Královéhradecký kraj
  - NEUROSPOL Sro, Havířov
  - Fakultni nemocnice v Motole, Prague
  - Krajska Zdravotni a.s. Nemocnice Teplice Oz, Teplice, Ústecký kraj
- France (7):
  - Hôpital Guillaume Et René Laënnec, Nantes, Loire-Atlantique
  - Hôpital Maison Blanche, Reims, Marne
  - Hôpital Roger Salengro, Lille, Nord
  - Hôpital Sud, Amiens, Somme
  - Hopital Gabriel Montpied, Clermont-Ferrand
  - CHRU Nancy, Nancy
  - Fondation Rothschild, Paris
- Hungary (4):
  - Szegedi Tudományegyetem Szent-Györgyi Albert Klinikai Központ, Szeged, Csongrád megye
  - Uzsoki Utcai Korhaz, Budapest
  - Jahn Ferenc Dél-Pesti Kórház és Rendelöintézet, Budapest
  - Pécsi Tudományegyetem, Pécs
- Italy (6):
  - Azienda Ospedaliera Universitaria San Martino, Genoa, Liguria
  - Ospedale San Raffaele S.r.l., Milan, Lombardy
  - Azienda Ospedaliera Spedali Civili di Brescia - Presidio Ospedaliero di Montichiari, Montichiari, Lombardy
  - Fondazione Istituto San Raffaele G. Giglio di Cefalù, Cefalù, Palermo
  - Azienda Ospedaliero Universitaria Policlinico-Vittorio Emanuele, Catania, Sicily
  - Azienda Ospedaliera S. Antonio Abate di Gallarate, Gallarate, Varese
- Netherlands (2):
  - Erasmus MC, Rotterdam, South Holland
  - Zuyderland Medisch Centrum, Sittard-Geleen
- Poland (11):
  - Centrum Neurologii K. Selmaj, Lódz, Lódzkie
  - Wojskowy Instytut Medyczny, Warsaw, Masovian Voivodeship
  - Novo-Med Zielinski i wsp. Sp.J., Katowice, Silesian Voivodeship
  - Pomorskie Centrum Traumatologii im. M. Kopernika w Gdansku, Gdansk
  - Regionalny Szpital Specjalistyczny im. dr Wladyslawa Bieganskiego, Grudziądz
  - M.A.- Lek A.M.Maciejowscy Spolka Cywilna, Katowice
  - Gabriela Klodowska-Duda Neuro-Care NZOZ Site Management Organization, Katowice
  - Neurologiczny NZOZ Centrum Leczenia SM Osrodek Badan Klinicznych Dr n. med. Hanka Hertmanowska, Plewiska
  - Niepubliczny Zaklad Opieki Zdrowotnej NEURO-KARD Ilkowski i Partnerzy Spolka Partnerska Lekarzy, Poznan
  - SPZOZ Wojewodzki Szpital Specjalistyczny w Rybniku, Rybnik
  - EUROMEDIS Sp. z o.o., Szczecin
- Russia (6):
  - Kaluga Regional Hospital, Kaluga
  - Republican Clinical Hospital For Rehabilitation Treatment, Kazan'
  - Krasnoyarsk State Medical Academy, Krasnoyarsk
  - Perm State Medical Academy, Perm
  - City Center of MS Treatment based on Saint-Petersburg City Clinical Hospital #31, Saint Petersburg
  - Regional Clinical Hospital #3, Volgograd
- Serbia (4):
  - Clinical Center of Serbia, Belgrade, Belgrade
  - Military Medical Academy, Belgrade
  - Clinical Center Kragujevac, Kragujevac
  - General Hospital Uzice, Užice
- Spain (8):
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona, Catalonia
  - Hospital Universitario Reina Sofia, Córdoba, Córdoba
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Hospital Clinico San Carlos, Madrid, Madrid, Communidad Delaware
  - Hospital Universitario Virgen Macarena, Seville, Sevilla
  - Hospital de Basurto Osakidetza, Bilbao, Vizcaya
  - Hospital General Carlos Haya, Málaga
- Queen's Medical Centre, Nottingham, Nottinghamshire, United Kingdom

REFERENCES:
- [Derived] Cadavid D, Mellion M, Hupperts R, Edwards KR, Calabresi PA, Drulovic J, Giovannoni G, Hartung HP, Arnold DL, Fisher E, Rudick R, Mi S, Chai Y, Li J, Zhang Y, Cheng W, Xu L, Zhu B, Green SM, Chang I, Deykin A, Sheikh SI; SYNERGY study investigators. Safety and efficacy of opicinumab in patients with relapsing multiple sclerosis (SYNERGY): a randomised, placebo-controlled, phase 2 trial. Lancet Neurol. 2019 Sep;18(9):845-856. doi: 10.1016/S1474-4422(19)30137-1. Epub 2019 Jul 5. PMID 31285147
- [Derived] Wilhelm H, Schabet M. The Diagnosis and Treatment of Optic Neuritis. Dtsch Arztebl Int. 2015 Sep 11;112(37):616-25; quiz 626. doi: 10.3238/arztebl.2015.0616. PMID 26396053

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 419 participants were randomized; 1 participant was not dosed.
Groups:
- Placebo: Placebo once every 4 weeks intravenous (IV) infusion up to Week 72.
  Avonex once-weekly intramuscular (IM) injection up to Week 84.
- BIIB033, 3 mg/kg: BIIB033 3 mg/kg once every 4 weeks IV infusion up to Week 72.
  Avonex once-weekly IM injection up to Week 84.
Period: Overall Study
Arm/Group | Placebo | BIIB033, 3 mg/kg | BIIB033, 10 mg/kg | BIIB033, 30 mg/kg | BIIB033, 100 mg/kg
Started | 93 | 45 | 95 | 94 | 92
Randomized and Dosed | 93 | 45 | 95 | 93 | 92
Completed | 73 | 40 | 84 | 68 | 69
Not Completed | 20 | 5 | 11 | 26 | 23
Not completed — Other | 2 | 1 | 1 | 3 | 1
Not completed — Death | 0 | 0 | 0 | 1 | 0
Not completed — Investigator Decision | 5 | 0 | 0 | 4 | 6
Not completed — Withdrawal by Subject | 9 | 2 | 6 | 8 | 8
Not completed — Lost to Follow-up | 0 | 0 | 0 | 2 | 1
Not completed — Adverse Event | 4 | 2 | 4 | 7 | 7
Not completed — Not Dosed | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population: all randomized participants who received at least 1 dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | BIIB033, 3 mg/kg | BIIB033, 10 mg/kg | BIIB033, 30 mg/kg | BIIB033, 100 mg/kg | Total
Number analyzed (Participants) | 93 | 45 | 95 | 93 | 92 | 418
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.5 (9.29) | 36.5 (9.47) | 40.5 (9.78) | 40.9 (9.70) | 39.8 (9.10) | 39.8 (9.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 24 | 59 | 61 | 66 | 277
  Male | 26 | 21 | 36 | 32 | 26 | 141

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Confirmed as Improvement Responders for Primary Multicomponent Endpoint
Description: Estimated proportion of participants experiencing confirmed improvement in any 1 or more of the following components: a ≥1 point decrease in the Expanded Disability Status Scale (EDSS) score from a baseline score of <=6.0 (decrease sustained for ≥3 months); a ≥15% improvement from baseline in time to complete 9-Hole Peg Test (9HPT) by either hand (improvement sustained for ≥3 months for the same hand), where the time is the average time of 2 trials per hand at the same visit; a ≥15% improvement from baseline in time to complete Timed 25-Foot Walk (T25FW) test (improvement sustained for ≥3 months), where the time is the average time of 2 trials at the same visit; or a ≥15% improvement from baseline 3-Second Paced Auditory Serial Addition Test (PASAT-3) score (improvement sustained for 3 months or greater). Estimated proportion of responders is based on logistic regression adjusted for multiple sclerosis (MS) type, region and baseline component assessments.
Time Frame: 72 weeks
Population: Intent-to-treat population: all randomized participants who received at least 1 dose of study treatment and included in the efficacy analysis (6 participants were excluded due to study site Good Clinical Practice deviation).
Measure: Number; unit: proportion of participants
Arm/Group | Placebo | BIIB033, 3 mg/kg | BIIB033, 10 mg/kg | BIIB033, 30 mg/kg | BIIB033, 100 mg/kg
Number analyzed (Participants) | 91 | 45 | 94 | 91 | 91
proportion of participants | 0.516 | 0.511 | 0.656 | 0.688 | 0.412
Statistical Analysis 1: Comparison: Placebo vs BIIB033, 3 mg/kg; Test type: Superiority or Other; p = 0.9584, Regression, Logistic; Odds ratios, 95% CI and p-values are based on logistic regression adjusted for MS type, region and baseline component assessments; Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.46 to 2.07]
Statistical Analysis 2: Comparison: Placebo vs BIIB033, 10 mg/kg; Test type: Superiority or Other; p = 0.0636, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.79, 95% CI 2-sided [0.97 to 3.31]
Statistical Analysis 3: Comparison: Placebo vs BIIB033, 30 mg/kg; Test type: Superiority or Other; p = 0.0220, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 2.06, 95% CI 2-sided [1.11 to 3.84]
Statistical Analysis 4: Comparison: Placebo vs BIIB033, 100 mg/kg; Test type: Superiority or Other; p = 0.1771, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.66, 95% CI 2-sided [0.36 to 1.21]
Statistical Analysis 5: Comparison: Placebo vs BIIB033, 3 mg/kg vs BIIB033, 10 mg/kg vs BIIB033, 30 mg/kg vs BIIB033, 100 mg/kg; Test type: Superiority or Other; p = 0.8931, Trend test; Trend test p-value is based on a linear contrast in logistic regression

2. Secondary Outcome: Proportion of Participants Confirmed as Worsening Responders for Primary Multicomponent Endpoint
Description: Estimated proportion of participants experiencing confirmed clinical worsening in 1 or more components of the multicomponent endpoint (EDSS, T25FW, 9HPT, or PASAT-3) over 72 weeks, defined as: a ≥1.0 point increase in EDSS from a baseline score of ≤5.5 or a ≥0.5 point increase from a baseline score equal to 6.0 (increase sustained for 3 months or greater); a ≥15%worsening from baseline in time to complete T25FW test (worsening sustained for 3 months or greater), where the time is the average of 2 trials at the same visit; a ≥15% worsening from baseline in time to complete 9HPT by either hand (worsening sustained for 3 months or greater for the same hand), where the time is the average of 2 trials for each hand at the same visit; a ≥15% worsening from baseline in PASAT-3 score (worsening sustained for 3 months or greater). Estimated proportion of responders is based on logistic regression adjusted for MS type, region and baseline component assessments.
Time Frame: 72 weeks
Population: as for outcome 1
Measure: Number; unit: proportion of participants
Arm/Group | Placebo | BIIB033, 3 mg/kg | BIIB033, 10 mg/kg | BIIB033, 30 mg/kg | BIIB033, 100 mg/kg
Number analyzed (Participants) | 91 | 45 | 94 | 91 | 91
proportion of participants | 0.403 | 0.304 | 0.509 | 0.489 | 0.369
Statistical Analysis 1: Comparison: Placebo vs BIIB033, 3 mg/kg; Test type: Superiority or Other; p = 0.3058, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.65, 95% CI 2-sided [0.28 to 1.49]
Statistical Analysis 2: Comparison: Placebo vs BIIB033, 10 mg/kg; Test type: Superiority or Other; p = 0.1873, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.53, 95% CI 2-sided [0.81 to 2.89]
Statistical Analysis 3: Comparison: Placebo vs BIIB033, 30 mg/kg; Test type: Superiority or Other; p = 0.2766, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.42, 95% CI 2-sided [0.76 to 2.65]
Statistical Analysis 4: Comparison: Placebo vs BIIB033, 100 mg/kg; Test type: Superiority or Other; p = 0.6578, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.86, 95% CI 2-sided [0.45 to 1.65]
Statistical Analysis 5: Comparison: Placebo vs BIIB033, 3 mg/kg vs BIIB033, 10 mg/kg vs BIIB033, 30 mg/kg vs BIIB033, 100 mg/kg; Test type: Superiority or Other; p = 0.5255, Trend test; Trend test p-value is based on a linear contrast in logistic regression

3. Secondary Outcome: Number of Participants Experiencing Adverse Events (AEs) and Serious Adverse Events (SAEs) and Discontinuations Due to AEs
Description: An AE was any untoward medical occurrence that did not necessarily have a causal relationship with this treatment. An SAE was any untoward medical occurrence that at any dose: resulted in death; in the view of the Investigators, placed the participant at immediate risk of death (a life-threatening event); however, this did not include an event that, had it occurred in a more severe form, might have caused death; required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; resulted in a congenital anomaly/birth defect; any other medically important event that, in the opinion of the Investigators, could have jeopardized the participant or may have required intervention to prevent one of the other outcomes listed in the definition above.
Time Frame: Up to 84 weeks
Population: Safety Population: all participants who received at least 1 dose of study treatment.
Measure: Number; unit: participants
Groups:
- BIIB033 Total: BIIB033 3, 10, 30, or 100 mg/kg once every 4 weeks IV infusion
Arm/Group | Placebo | BIIB033, 3 mg/kg | BIIB033, 10 mg/kg | BIIB033, 30 mg/kg | BIIB033, 100 mg/kg | BIIB033 Total
Number analyzed (Participants) | 93 | 45 | 95 | 93 | 92 | 325
participants
  Any event | 79 | 39 | 84 | 79 | 73 | 275
  Moderate or severe event | 59 | 26 | 59 | 59 | 58 | 202
  Severe event | 7 | 2 | 6 | 6 | 7 | 21
  BIIB033/placebo-related event | 8 | 8 | 15 | 12 | 16 | 51
  Avonex-related event | 51 | 28 | 58 | 54 | 50 | 190
  Serious event | 13 | 4 | 11 | 20 | 16 | 51
  BIIB033/placebo-related serious event | 1 | 0 | 0 | 1 | 5 | 6
  Avonex-related serious event | 1 | 0 | 0 | 2 | 1 | 3
  Event leading to discontinuation of treatment | 4 | 2 | 3 | 7 | 8 | 20
  Event leading to withdrawal from study | 4 | 2 | 4 | 8 | 7 | 21

4. Secondary Outcome: Pharmacokinetics: BIIB033 Plasma Concentrations up to Week 84
Time Frame: Up to 84 weeks
Population: PK Population: participants who received at least 1 dose of BIIB033 and had at least 1 serum concentration data point on record.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | BIIB033, 3 mg/kg | BIIB033, 10 mg/kg | BIIB033, 30 mg/kg | BIIB033, 100 mg/kg
Number analyzed (Participants) | 45 | 95 | 92 | 92
µg/mL
  Baseline, predose; n=44, 95, 92, 92 | 0.00 (0.00) | 0.01 (0.13) | 7.79 (74.75) | 0.42 (4.07)
  Baseline, postdose; n=44, 95, 91, 92 | 66.70 (16.00) | 244.76 (77.90) | 688.47 (245.73) | 2298.20 (712.91)
  Week 4, predose; n=45, 93, 91, 88 | 10.82 (4.11) | 46.28 (33.15) | 138.54 (92.82) | 457.96 (308.09)
  Week 4, postdose; n=45, 94, 89, 85 | 123.96 (315.66) | 279.67 (100.01) | 784.08 (204.31) | 2763.26 (823.42)
  Week 8, predose; n=45, 95, 89, 85 | 23.55 (54.96) | 65.48 (52.53) | 195.29 (118.24) | 603.11 (425.58)
  Week 8, postdose; n=44, 94, 88, 79 | 86.29 (52.74) | 294.44 (78.61) | 861.60 (274.56) | 2751.25 (697.42)
  Week 16, predose; n=43, 94, 86, 79 | 19.96 (9.74) | 71.80 (25.13) | 231.94 (125.42) | 695.11 (438.57)
  Week 16, postdose; n=41, 93, 85, 78 | 85.95 (29.04) | 309.38 (83.38) | 881.45 (211.32) | 2921.09 (1118.88)
  Week 24, predose; n=42, 93, 85, 74 | 36.41 (85.48) | 77.88 (33.68) | 230.46 (77.40) | 699.63 (400.49)
  Week 24, postdose; n=42, 92, 82, 76 | 144.12 (373.36) | 318.01 (84.74) | 940.29 (231.35) | 2870.29 (874.28)
  Week 36, predose; n=41, 88, 79, 74 | 25.33 (18.28) | 85.05 (44.67) | 238.48 (73.75) | 725.22 (344.01)
  Week 36, postdose; n=42, 88, 77, 73 | 94.62 (21.89) | 339.17 (88.96) | 197.86 (197.96) | 3048.66 (989.34)
  Week 48, predose; n=39, 85, 74, 70 | 20.78 (6.26) | 80.28 (31.62) | 272.88 (167.79) | 806.70 (541.78)
  Week 48, postdose; n=42, 85, 75, 72 | 90.07 (23.37) | 334.12 (78.43) | 955.25 (193.34) | 3167.07 (1144.25)
  Week 60, predose; n=41, 84, 70, 68 | 21.29 (12.34) | 81.77 (30.24) | 243.18 (78.57) | 694.12 (200.41)
  Week 60, postdose; n=42, 84, 71, 71 | 93.11 (35.98) | 335.10 (93.29) | 939.17 (255.64) | 3330.70 (1076.88)
  Week 72, predose; n=41, 85, 72, 68 | 19.53 (9.34) | 78.94 (29.95) | 215.09 (62.98) | 819.39 (577.60)
  Week 72, postdose; n=38, 84, 69, 68 | 82.96 (31.84) | 313.13 (87.22) | 868.39 (231.14) | 3145.82 (1233.66)
  Week 84; n=40, 81, 69, 69 | 2.44 (1.25) | 12.77 (6.80) | 46.16 (31.52) | 127.69 (65.46)

ADVERSE EVENTS:
Time Frame: From first dosing of study treatment through end of study (Week 84)
Groups:
- BIIB033 3 mg/kg: BIIB033 3 mg/kg once every 4 weeks IV infusion
- BIIB033 10 mg/kg: BIIB033 10 mg/kg once every 4 weeks IV infusion
- BIIB033 30 mg/kg: BIIB033 30 mg/kg once every 4 weeks IV infusion
- BIIB033 100 mg/kg: BIIB033 100 mg/kg once every 4 weeks IV infusion
Arm/Group | Placebo | BIIB033 3 mg/kg | BIIB033 10 mg/kg | BIIB033 30 mg/kg | BIIB033 100 mg/kg
Serious Adverse Events (participants affected / at risk) | 13/93 | 4/45 | 11/95 | 20/93 | 16/92
Other Adverse Events (participants affected / at risk) | 74/93 | 38/45 | 79/95 | 70/93 | 67/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=93) | BIIB033 3 mg/kg (N=45) | BIIB033 10 mg/kg (N=95) | BIIB033 30 mg/kg (N=93) | BIIB033 100 mg/kg (N=92)
Hypochromic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 4
Cystitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 0 | 0 | 0 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Multiple sclerosis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Multiple sclerosis relapse (Nervous system disorders) | 7 | 2 | 6 | 10 | 6
Radicular syndrome (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Secondary progressive multiple sclerosis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Trigeminal neuralgia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Acute psychosis (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Bipolar I disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Uterine polyp (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=93) | BIIB033 3 mg/kg (N=45) | BIIB033 10 mg/kg (N=95) | BIIB033 30 mg/kg (N=93) | BIIB033 100 mg/kg (N=92)
Diarrhoea (Gastrointestinal disorders) | 3 | 5 | 3 | 3 | 3
Asthenia (General disorders) | 8 | 1 | 5 | 6 | 3
Chills (General disorders) | 5 | 4 | 4 | 8 | 4
Fatigue (General disorders) | 8 | 6 | 5 | 7 | 7
Influenza like illness (General disorders) | 37 | 17 | 51 | 34 | 38
Pyrexia (General disorders) | 7 | 9 | 8 | 12 | 11
Influenza (Infections and infestations) | 4 | 3 | 6 | 4 | 6
Nasopharyngitis (Infections and infestations) | 16 | 3 | 12 | 8 | 10
Pharyngitis (Infections and infestations) | 2 | 5 | 4 | 3 | 3
Sinusitis (Infections and infestations) | 5 | 2 | 2 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 13 | 4 | 21 | 11 | 9
Urinary tract infection (Infections and infestations) | 12 | 7 | 14 | 9 | 13
Fall (Injury, poisoning and procedural complications) | 10 | 0 | 4 | 8 | 5
Alanine aminotransferase increased (Investigations) | 3 | 2 | 5 | 6 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 2 | 4 | 7 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 3 | 9 | 6 | 6
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 3 | 2 | 2 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 1 | 2 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 1 | 5 | 4 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 5 | 5 | 7 | 1
Headache (Nervous system disorders) | 23 | 8 | 19 | 13 | 11
Multiple sclerosis relapse (Nervous system disorders) | 30 | 17 | 35 | 36 | 28
Anxiety (Psychiatric disorders) | 4 | 0 | 5 | 2 | 3
Depressed mood (Psychiatric disorders) | 2 | 3 | 1 | 2 | 1
Depression (Psychiatric disorders) | 6 | 2 | 6 | 7 | 2
Insomnia (Psychiatric disorders) | 1 | 2 | 4 | 6 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.